CLINICAL TRIAL: NCT06150768
Title: Biting Force and Quality of Life in Porcelain-fused-to Metal Versus Zirconia Implant- Supported in Mandibular Kennedy Class II ( In Vivo Study )
Brief Title: Porcelain-fused-to-metal Versus Zirconia Implant- Supported in Mandibular Kennedy Class II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RecIM 092305
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Partial Edentulism Class II; Dental Implants; Implant
Keywords: Dental Implants; Edentulous; partially; dental prosthesis; implant-supported; fixed partial denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Intervention Model Description: Control group (1) will receive a CoCr removable partial denture; in the other two groups (2) and (3), implants will be inserted to restore missed posterior teeth (second mandibular premolar and second mandibular molar) in the span area using a two-stage surgical technique with the help of a radiographic and surgical stent. After a three-month osseointegration period, implants will be loaded with three units of anatomical PFM fixed partial dentures in group (2), while in group (3), implants will be loaded with three units of anatomical Zirconia fixed partial dentures. Biting force will be measured using a biting force sensor for both the intact and restored sides at the time of delivery of the removable partial denture and at loading of implants, after 2, 4, and 6 months. Patient satisfaction will be assessed through a quality-of-life questionnaire at the recall appointments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group Cobalt Chromium Removable Partial Denture (Active Comparator): The patient will receive a Cobalt Chromium Removable Partial Denture to restore missing posterior teeth in Kennedy Class II cases. The denture will be fabricated by conventional lost-wax and processing techniques.
  Interventions: Device: Cobalt Chromium Removable Partial Denture
- Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture (Experimental): Two dental implants will be placed to restore missed posterior teeth (second mandibular premolar and second mandibular molar) in Kennedy Class II cases by using a two-stage surgical technique with the help of a radiographic and surgical stent. After a three-month osseointegration period, implants will be loaded with three units of anatomical Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture
  Interventions: Device: Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture
- Implant-Supported Zirconia fixed partial denture (Experimental): Two dental implants will be placed to restore missed posterior teeth (second mandibular premolar and second mandibular molar) in Kennedy Class II cases by using a two-stage surgical technique with the help of a radiographic and surgical stent. After a three-month osseointegration period, implants will be loaded with three units of anatomical implant-supported Zirconia fixed partial dentures
  Interventions: Device: Implant-Supported Zirconia Fixed Partial Denture.

INTERVENTIONS:
Device: Cobalt Chromium Removable Partial Denture — The patient will receive Removable Partial Denture to restore missing teeth in Kennedy Class II cases.
  Other Names: Combined Removable Partial denture.
  Arms: Control group Cobalt Chromium Removable Partial Denture
Device: Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture — The patient will receive Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture to restore missing teeth in Kennedy Class II cases.
  Other Names: : Implant-Supported Porcelain-Fused-to-Metal-Fixed bridge
  Arms: Implant-Supported Porcelain-Fused-to-Metal-Fixed Partial Denture
Device: Implant-Supported Zirconia Fixed Partial Denture. — The patient will receive Implant-Supported Zirconia Fixed Partial Denture to restore missing teeth in Kennedy Class II cases.
  Other Names: Implant-Supported Zirconia Fixed bridge.
  Arms: Implant-Supported Zirconia fixed partial denture

SUMMARY:
The goal of this randomized clinical trial is to compare biting force and patient satisfaction in three groups. Patients in the control group number one will receive a CoCr removable partial denture, and in the other two groups, implants will be inserted to restore missed posterior teeth (second mandibular premolar and second mandibular molar) in the span area. After three months, implants will be loaded with three units of anatomical PFM-fixed partial dentures in group number two, while in group number three, implants will be loaded with three units of anatomical Zirconia-fixed partial dentures. Biting force will be measured bilaterally at the time of delivery of the removable partial denture and delivery of fixed partial dentures after two, four, and six months. Patient satisfaction will be assessed through a quality-of life questionnaire at the six-months recall appointment

DETAILED DESCRIPTION:
Thirty-three partially edentulous patients will be recruited. Patients will be randomly divided into three groups. Patients in the control group number one will receive a CoCr removable partial denture; in the other two groups, implants will be inserted to restore missed posterior teeth (second mandibular premolar and second mandibular molar) in the span area using a two-stage surgical technique with the help of a radiographic and surgical stent. Pre-surgical and post-surgical prescription of antibiotics, anti-inflammatory drugs, analgesic drugs, and mouthwash for one week, then a follow-up will be done at the suture removal appointment. After a three-month osseointegration period, implants will be loaded with three units of anatomical PFM-fixed partial dentures in group number two, while in group number three, implants will be loaded with three units of anatomical Zirconia-fixed partial dentures. Recall appointments will be scheduled for the patients two, four, and six months after loading for the collection of the data. Biting force will be measured using a biting force sensor for both the intact and restored sides at the time of delivery of the removable partial denture and at the loading of implants after two, four, and six months. Patient satisfaction will be assessed through a quality-of-life questionnaire at the six-months recall appointment.

ELIGIBILITY:
Inclusion Criteria:

* Kennedy Class II mandibular arch where the last standing abutment is the first premolar, opposed by a fully dentate maxilla (either natural dentition or fixed prostheses).
* A minimum of 12 millimeters of bone height above the inferior alveolar canal diagnosed from the pre-operative cone beam CT.
* Sufficient inter-arch space to accommodate the implant supported fixed partial denture.

Exclusion Criteria:

* Patients with bone or mucosal diseases.
* Heavy smokers.
* Patients with uncontrolled metabolic disorders such as diabetes mellitus.
* Patients with parafunctional habits.
* Patients with conditions that might complicate the treatment, such as: severe gag reflex, limited mouth opening.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of biting force | Biting force will be measured by newtons unit per minute using a biting force sensor for both the intact and restored sides at the time of delivery of the removable partial denture ( baseline ) and at loading of implants, after 2, 4, and 6 months.
  improvement of Biting force in two different implants supported partial dentures.

SECONDARY OUTCOMES:
Oral health-related quality of life ( OHRQoL ) Measurement | At the time of delivery of the removable partial denture ( baseline ) and at loading of implants, after 2, 4, and 6 months. Patient satisfaction will be assessed through a quality-of-life questionnaire at the recall appointments.
  OHRQoL was measured by using the original version of the Oral Health Impact Profile OHIP-14, which has been shown to be valid and reliable. The questionnaire included sevendomains-functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap-with two questions each.
  For each item responses were never, hardly ever, occasionally, fairly often and very often.
  Items were scored on a 5-point scale ranging from 0 (never), to 1 (hardly ever), 2 (occasionally), 3 (fairly often) and 4 (very often)

CONTACTS AND LOCATIONS:
Overall Officials: Ingy T Lebshtien, PHD, Study Director — Faculty of Dentistry Ain Shams University; Noha M El Hussieny, PHD, Principal Investigator — Faculty of Dentistry Ain Shams University; Omnia MS Refai, PHD, Principal Investigator — Faculty of Dentistry Ain Shams University; Ali M Fouda, Principal Investigator — Faculty of Dentistry Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD that will be published will include the patients' gender, age and the outcome results without disclosing any personal data of the individuals.
Supporting Information: Study Protocol
Time Frame: The IPD will be available after the end of the study, and it will be available for 12 months after the publication date of the study.

REFERENCES:
- [Background] Bandiaky ON, Lokossou DL, Soueidan A, Le Bars P, Gueye M, Mbodj EB, Le Guehennec L. Implant-supported removable partial dentures compared to conventional dentures: A systematic review and meta-analysis of quality of life, patient satisfaction, and biomechanical complications. Clin Exp Dent Res. 2022 Feb;8(1):294-312. doi: 10.1002/cre2.521. Epub 2022 Jan 11. PMID 35014207
- [Background] Bural C, Buzbas B, Ozatik S, Bayraktar G, Emes Y. Distal extension mandibular removable partial denture with implant support. Eur J Dent. 2016 Oct-Dec;10(4):566-570. doi: 10.4103/1305-7456.195180. PMID 28042277
- [Background] Behr M, Zeman F, Passauer T, Koller M, Hahnel S, Buergers R, Lang R, Handel G, Kolbeck C. Clinical performance of cast clasp-retained removable partial dentures: a retrospective study. Int J Prosthodont. 2012 Mar-Apr;25(2):138-44. PMID 22371834
- [Background] Erkmen E, Meric G, Kurt A, Tunc Y, Eser A. Biomechanical comparison of implant retained fixed partial dentures with fiber reinforced composite versus conventional metal frameworks: a 3D FEA study. J Mech Behav Biomed Mater. 2011 Jan;4(1):107-16. doi: 10.1016/j.jmbbm.2010.09.011. Epub 2010 Oct 1. PMID 21094484
- [Background] Nazari V, Ghodsi S, Alikhasi M, Sahebi M, Shamshiri AR. Fracture Strength of Three-Unit Implant Supported Fixed Partial Dentures with Excessive Crown Height Fabricated from Different Materials. J Dent (Tehran). 2016 Nov;13(6):400-406. PMID 28243301
- [Background] Gokcen-Rohlig B, Saruhanoglu A, Cifter ED, Evlioglu G. Applicability of zirconia dental prostheses for metal allergy patients. Int J Prosthodont. 2010 Nov-Dec;23(6):562-5. PMID 21209994
- [Background] Pelaez J, Cogolludo PG, Serrano B, Serrano JF, Suarez MJ. A four-year prospective clinical evaluation of zirconia and metal-ceramic posterior fixed dental prostheses. Int J Prosthodont. 2012 Sep-Oct;25(5):451-8. PMID 22930766
- [Background] Gu Y, Bai Y, Xie X. Bite Force Transducers and Measurement Devices. Front Bioeng Biotechnol. 2021 Apr 9;9:665081. doi: 10.3389/fbioe.2021.665081. eCollection 2021. PMID 33898409